CLINICAL TRIAL: NCT03560934
Title: Effect of Tetrahydrocannabinol (THC) on Sleep in Humans
Brief Title: Tetrahydrocannabinol (THC) and Sleep
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Nicole Bowles, Assistant Professor, Oregon Institute of Occupational Health Sciences, Oregon Health and Science University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00018052
Record Dates: First submitted 2018-02-09; First posted 2018-06-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-06

CONDITIONS: Sleep; THC; Marijuana; Cannabis
MeSH Terms: conditions — Marijuana Abuse | interventions — Dronabinol

STUDY DESIGN:
Intervention Model Description: Participants are initially categorized as non-frequent or frequent cannabis users based on their cannabis use behavior and then receive the same treatment of 10-60mg dronabinol upon participation in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Frequent Cannabis Users (Experimental): Subjects categorized as frequent cannabis users (>3x/week for 3 months) will receive a single dose of 10-60mg dronabinol on the second or third night of their stay in the clinical laboratory, one hour prior to bedtime and five minutes after completion of a study snack. The other night, participants will receive a placebo.
  Dronabinol is an orally active, synthetic THC currently indicated for weight loss in patients with acquired immune deficiency syndrome (AIDS) or anorexia and for nausea and vomiting associated with cancer. Dronabinol is nearly absorbed (90%-95%) after a single oral dose of the capsule formulation with 10-20% of the administered dose researching the systemic circulation due to extensive first-pass hepatic metabolism and high lipid solubility. The onset of action is ~30 to 60 minutes with peak effects from 2-4-h following dose (Fig. 2) (34). The 10-60mg of dronabinol will be administered by OHSU's research pharmacy services.
  Interventions: Drug: Dronabinol
- Non Cannabis Users (Experimental): Non-cannabis users (who have not used cannabis more than 10 times in their lifetime) will undergo the same single dose dronabinol and placebo as the frequent cannabis user arm, under the identical study procedure.
  Interventions: Drug: Dronabinol

INTERVENTIONS:
Drug: Dronabinol — Single dose oral administration of 10-60mg dronabinol prior to night 2 or 3 sleep in the clinical laboratory.
  Other Names: Marinol

SUMMARY:
The investigators will test the effects of 10-60mg dronabinol (oral THC) on sleep in non-frequent and frequent cannabis users.

DETAILED DESCRIPTION:
The investigators plan to test the effects of 10-60 mg dronabinol (oral THC) on subjective (surveys) and objective (polysomnographically scored (PSG)) sleep in non-frequent and frequent cannabis users following an acclimation and baseline night of sleep. The mornings after baseline sleep and dronabinol administration, cognitive performance will also be measured and participants may also perform morning typical behaviors such as change in posture (getting out of bed/tilt test) and mild intensity physical activity. This pilot study is in healthy young adults without a history of chronic disease.

ELIGIBILITY:
Inclusion Criteria:

* Frequent Cannabis Use (>3x/week for the prior 3 months) or
* No Cannabis Use (Less than 10x ever)

Exclusion Criteria:

* Sleep Apnea
* Pregnancy
* Diabetes
* Cardiovascular disease
* Chronic Pain
* History of seizures
* Severe Hepatic impairment
* Conditions associated with clinically relevant cognitive impairment
* Symptoms of acute or active illness (e.g., fever and leukocytosis)
* Evidence of psychopathology on the Beck Depression Index II (BDI-II or in a structured clinical interview with a physician
* History of severe psychiatric illnesses (including such as alcoholism, drug dependency including a cannabis use disorder score ≥12 on the Cannabis Use Disorders Identification Test (CUDIT) (28) or >1 withdrawal symptom on the Marijuana Withdrawal Checklist (MWC (29)) , major depression, manic depressive illness, schizophrenic disorders, panic disorder, generalized anxiety disorder, post-traumatic stress disorder, agoraphobia, claustrophobia, paranoid personality disorder, schizoid personality disorder, schizotypal personality disorder, borderline personality disorder, and antisocial personality disorder.)
* History of having been treated with antidepressants, neuroleptic medications, or tranquilizers.
* Volunteers must be drug-free (including caffeine, nicotine, alcohol and herbal medications) for the duration of the screening and study period (with the exception of THC), with no dependence on drugs (e.g. cocaine, opioids, amphetamine, methamphetamine, PCP, benzodiazepines, barbiturates, methadone, MDMA); or alcohol dependency.
* Current Nicotine use ( or history of more than 5 'pack years' of smoking)
* Current use of prescription or over the counter medications
* History of shift work in the last 6 months
* Travel across >2 time zones during the month prior to the study
* Habitual bedtime after 1am or waketime before 5am

Ages: 21 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-09-19 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Sleep Stages | Over the 3-night stay.
  Polysomnographic recordings will be measured and scored across the three sleep periods for timing and sleep stages.
Psychomotor Vigilance Change Across Four Day Inpatient Stay | Over the 3-night stay.
  Psychomotor vigilance response times (in milliseconds) will be measured shortly after awakening each test morning.
Mean Change in Response Accuracy for Paced Auditory Serial Addition Test Across Four Day Inpatient Stay | Over the 3-night stay.
  Processing speed and working memory (response accuracy) will be measured shortly after awakening each test morning. Scores can range from a minimum of 0 to 60 correct responses with each test.
Mean Change in Response Accuracy for Word Recall Across Four Day Inpatient Stay | Over the 3-night stay.
  Verbal memory will be measured shortly after awakening each test morning. Scores can range from recalling 0 words to the complete list. Participants are blinded as to list length.
Mean changes in Intoxication Levels on the Visual Analog Scale | Over the 3-night stay.
  Assessed by visual analog scale (Minimum=0, Maximum=100). 0 is "Not at all" and 100 is "Extremely". Questions ask about feeling drug effect, high right now, and wanting more of the study drug.
Blood pressure | Over the 3-night stay.
  Blood pressure (BP) will be measured every 30 min during wake and every 15 minutes during sleep. Beat-by-beat (BP) will be measured during sleep using a non-invasive device employing the volume-clamp method with hydrostatic correction (BMeye Nexfin or AD Instruments NIBP). Additionally an automated calibrated sphygmomanometer will be used to record sporadic BP at intervals during an exercise challenge.
Heart Rate | Over the 3-night stay.
  For the duration of the study, 2 channels of EKG are recorded (RA-V6) and stored at a sample frequency of 256 Hz. This software will be used for peak detection (R-wave detection and subsequent heart rate variability (HRV) analysis to estimate cardiac vagal tone).
Endothelial Function | Over the 3-night stay.
  Endothelial Function will be measured as Flow Mediated Dilation in the brachial artery 10 minutes after each awakening and 20 minutes before each sleep period.

SECONDARY OUTCOMES:
Subjective measures of sleepiness/alertness | Over the 3-night stay.
  Subjective sleepiness and alertness will be measured regularly (~1/h) across wake periods during the study protocol using the Stanford Sleepiness Scale. The scale measures subjective sleepiness on a 1-5 point Likert scale with 5 indicating the highest degree of sleepiness and 1 indicating the lowest degree of sleepiness.
Caloric Intake | Over the 3-night stay.
  Participants will use a meal logging app to log all meals and beverages consumed for caloric/nutritional content and timing for a period prior to coming into the clinical laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Shea, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No